CLINICAL TRIAL: NCT04033380
Title: Clinical Efficacy of Ceramic vs Resin Bloc Endocrowns: Study Protocol for the Randomized Clinical Trial
Brief Title: Clinical Efficacy of Ceramic vs Resin Block Endocrown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NanFangH
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Tooth Diseases
Keywords: Ceramic, Resin Bloc, Endocrown , Root Canal Treatment, Molar
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin bloc endocrown (Active Comparator): composite-based blocs (Grandio Blocs, VOCO)
  Interventions: Device: Resin blocs (Grandio Blocs, VOCO)
- Ceramic endocrown (Active Comparator): glass ceramic zirconia enhanced lithium silicate glass ceramics (Suprinity, VITA)
  Interventions: Device: Ceramic (Suprinity, VITA)

INTERVENTIONS:
Device: Resin blocs (Grandio Blocs, VOCO) — composite-base bloc (Grandio Blocs, VOCO)
  Arms: Resin bloc endocrown
Device: Ceramic (Suprinity, VITA) — glass ceramic zirconia enhanced lithium silicate glass ceramics (Suprinity, VITA)
  Arms: Ceramic endocrown

SUMMARY:
Compare the comfort and durability of Ceramic (VITA,Suprinity ,VS) vs Resin Bloc (VOCO, Grandio Bloc,GB) Endocrown by chairside CAD/CAM system (computer aided design / manufacture).

Objective:To provide information of material selection for the chair-side restoration of the teeth after root canal treatment.

DETAILED DESCRIPTION:
Pulpal and periapical diseases are the main causes of tooth loss. Root canal treatment (RCT) is the only effective way to treat these diseases. However, failure of RCT is commonly seen without coronal restoration.Endocrown is a new type of onlay with a retainer in the pulp cavity which consists of a cervical margin in the form of a butt joint and a preparation of the pulp chamber.This restoration method is not only good at the preservation of residual tooth tissue, but also suitable for severely damaged molars or premolars after dental pulp treatment.More and more endondontist tend to use this ways because they are a minimally invasive solution in such cases.Endocrown is mainly made of glass-ceramics, which has the advantages of beautiful appearance, high hardness and good biocompatibility. However, ceramic materials are brittle and fracturable, and need to be sintered twice in the manufacturing process, which is relatively complex and time-consuming. Composite resin block material is a new type of composite material developed in recent years. It is used for chairside CAD/CAM restoration,It has beautiful and natural color, and its elastic modulus is close to dentin. Therefore, it is more compatible with natural teeth in performance.Moreover, In the process of making, the steps of secondary sintering and glazing are omitted and shortened. But, there was no sufficient data to verify which material was more effective. The main aim of this trial is to compare the clinical efficacy of ceramic vs resin-based bloc endocrown. Other objectives include looking for the prognostic and influence factors of the related effects.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is healthy and is 18-75 years old and has molar teeth and tooth root apex without evident damage and no root fracture, as determined by x-ray.
2. The patient has three or four walls of intact tooth tissue after root canal treatment
3. The patient has good oral hygiene.
4. The patient has signed an informed consent form.
5. The patient is not participating in any other clinical trial.
6. The patient has received a class A assessment according to FDI criteria for marginal adaptation after restoration.

Exclusion Criteria:

1. Obvious destruction of the apical tissue or presence of large cysts or both
2. Severe periodontitis
3. Oral malignant tumor(s)
4. Undergoing radiotherapy
5. Pregnancy
6. Mental illness or systemic diseases
7. Incapable of self-care
8. Unsuitable for the trial as deemed by the researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Marginal Adaptation | 2 years
  FDI criteria for dental restorations assessment（2010） This criteria is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as The overall score of the restoration, thus resulting in a single (ordinal) primary outcome.

SECONDARY OUTCOMES:
Fracture of material and retention： | 2 years
  Clinical evaluations were performed at baseline and 24 months according to FDI criteria by 2 independent evaluators. A: Intact; B: Crack apparent on transillumination; C: Fracture observable; D: Endocrown lost (state at which interface debond occurred).
wear | 2 years
  Clinical evaluations were performed at baseline and 24 months according to FDI criteria by 2 independent evaluators.
Recurrence of caries | 2 years
  Clinical evaluations were performed at baseline and 24 months according to FDI criteria by 2 independent evaluators.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjuan Yan, PHD, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- NanFang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997
- [Background] Marquillier T, Domejean S, Le Clerc J, Chemla F, Gritsch K, Maurin JC, Millet P, Perard M, Grosgogeat B, Dursun E. The use of FDI criteria in clinical trials on direct dental restorations: A scoping review. J Dent. 2018 Jan;68:1-9. doi: 10.1016/j.jdent.2017.10.007. Epub 2017 Oct 18. PMID 29055692
- [Derived] Wang J, Ling Z, Zheng Z, Zheng C, Gai Y, Zeng Y, Zhu X, Chen L, Wu B, Yan W. Clinical efficacy of ceramic versus resin-based composite endocrowns in Chinese adults: study protocol for a randomized controlled trial. Trials. 2020 Jun 22;21(1):559. doi: 10.1186/s13063-020-04506-9. PMID 32571397